CLINICAL TRIAL: NCT03085576
Title: National Tunisian Registry of Atrial Fibrillation
Acronym: NATURE-AF
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne de Cardiologie & de Chirurgie Cardio-Vasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-001-NATUREAF
Record Dates: First submitted 2017-03-05; First posted 2017-03-21 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Anticoagulation; Stroke; Vitamin K antagonist; Cardioversion; INR (International Normalized Ratio)
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A non-interventional, national longitudinal study of atrial fibrillation performed with 91 cardiologists.

DETAILED DESCRIPTION:
The NATURE-AF study is carried out in Tunisia at cardiology consultations in hospitals and in the liberal sector. A total of 91 cardiologists participate in the selection of patients as investigators. The study is a longitudinal non-interventional registry of atrial fibrillation. The data collected are managed by the DACIMA Clinical Suite® platform, which complies with international standards: FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPPA (Health Insurance Portability and Accountability Act), ICH (International Conference on Harmonisation), MedDRA (Medical Dictionary for Regulatory Activities). The DACIMA Clinical Suite® platform allows to track the data entered, check for inconsistencies and missing data, and schedule monitoring visits. A Steering Committee is set up to monitor patient inclusions, verify data sources, perform audit trails and prepare the statistical analysis plan for the study.

ELIGIBILITY:
Inclusion Criteria:

* At least one episode of atrial fibrillation, documented on a 12-lead ECG and / or a rhythmic holter (duration of the episode: 30 seconds or more)
* Recent atrial fibrillation diagnosed for less than a year
* Regular monitoring every 3 months is ensured
* Informed, read and signed consent

Exclusion Criteria:

* Estimated life expectancy at less than 12 months
* Transient atrial fibrillation due to reversible cause (eg acute myocardial infarction, following cardiac surgery, acute alcohol intoxication, hyperthyroidism, pulmonary embolism or other acute pulmonary disease, pericarditis, myocarditis, hydro-electrolyte disorder, metabolic disorder)
* Cardiac surgery ≤ 3 months
* Atrial flutter isolated without atrial fibrillation
* Mental disorders
* Ongoing anticoagulation for reasons other than atrial fibrillation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke or transient ischemic attack, thromboembolic events and cardiovascular death | Every 3 months up to 1 year
  Number of patients with ischemic stroke and/or transient ischemic attack, and/or arterial embolization during the follow-up period

SECONDARY OUTCOMES:
Haemorrhagic accidents | Every 3 months up to 1 year
  All bleeding events (digestive, cerebral, other locations)
Measurement of INR (International Normalized Ratio) | Every month for 1 year
  INR measurement of venous blood sampling
TTR (percent Time in Therapeutic INR Range) | 1 year
  The mean TTR obtained in patients who received anticoagulant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Faouzi Addad, Professor, Study Chair — Société Tunisienne de Cardiologie et de Chirurgie Cardiovasculaire
Locations (1):
- STCCCV - Société Tunisienne de Cardiologie et de Chirurgie Cardio-Vasculaire, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben Halima A, Ouali S, Mourali MS, Chabrak S, Chettaoui R, Ben Halima M, Haggui A, Larbi N, Krichene S, Marrakchi S, Kacem S, Chrigui R, Abbes MF, Baccar H, Baraket N, Ben Halima N, Ben Khalfallah A, Ben Mbarek M, Ben Youssef S, Boughzala E, Boujnah MR, Drissa H, Gamra H, Gasmi A, Haouala H, Harrath Y, Issa I, Jeridi G, Kachboura S, Kammoun S, Kraiem S, Maatouk F, Milouchi S, Nasraoui W, Neji A, Sayahi K, Sdiri W, Smati W, Tlili S, Abid L, Abdesselem S, Zakhama L, Mahdhaoui A, Kammoun H, Ben Omrane S, Addad F. Design and Rationale of the National Tunisian Registry of Atrial Fibrillation: Protocol for a Prospective, Multicenter Trial. JMIR Res Protoc. 2018 Oct 15;7(10):e181. doi: 10.2196/resprot.8523. PMID 30322836
- [Background] Ouali S, Ben Halima A, Chabrak S, Chettaoui R, Ben Halima M, Haggui A, Krichane S, Noureddine L, Marrakchi S, Charfeddine S, Hassine M, Sayahi K, Abbes Mohamed F, Nasraoui W, Ajmi H, Ben Miled M, Jebbari Z, Meghaieth MA, Allouche E, Mechmeche R, Zakhama L, Sdiri W, Ben Khalfallah A, Gharbi A, Milouchi S, Neji A, Antit S, Battikh K, Drissa M, Kaabachi S, Najar T, Tlili R, Chahbani I, Charfeddine H, Ben MM, Braham S, Maatouk F, Abdesselem S, Ayari M, Garbaa R, Hamrouni N, Mbarek D, Rekik H, Zaghdoudi H, Ayadi W, Baraket F, Ben Brahim K, Ben Romdhane M, Bousadia H, Brahim W, Mezri M, Guesmi A, Ounissi T, Kammoun S, Smati W, Tlili S, Zoughi K, Zemni J, Cheikh Bouhlel M, Islem S, Jemli R, Joulak A, Mzoughi K, Naanea H, Hached L, Hadrich M, Hmem M, Kacem S, Kammoun I, Othmani R, Ouerghi A, Abid S, Ennouri R, Haidar S, Heraiech S, Jammali M, Jarrar M, Riahi L, Trimech B, Azaiez MA, Azzouzi F, Ben Jemaa K, Ben Rejab O, Chrigui R, Wechtati W, Boughzela E, Jridi G, Bezdah L, Kraiem S, Drissa H, Ben Youssef S, Fehri W, Kachboura S, Gamra H, Kammoun S, Mourali MS, Addad F, Abid L. Epidemiological characteristics, management, and outcomes of atrial fibrillation in TUNISIA: Results from the National Tunisian Registry of Atrial Fibrillation (NATURE-AF). Clin Cardiol. 2021 Apr;44(4):501-510. doi: 10.1002/clc.23558. Epub 2021 Mar 11. PMID 33704830
- See also: Medscape : A first register on AF in the Maghreb — https://francais.staging.medscape.com/voirarticle/3606891?fbclid=IwAR1CgOQVZhdvIgVnI-ENiCMDIYgc2x22NF7GFcdj7_rADztgmccRwc6Stgc